CLINICAL TRIAL: NCT04792827
Title: Feasibility of a Fast Track Concept for Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation Based on Individualized Low-dose Analgosedation and Preprocedural Fluid Optimization Using Echocardiography.
Brief Title: Fast Track Concept for Transfemoral TAVI
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Prof. Dr. med. Jochen Renner, University Hospital Schleswig-Holstein
Other Study IDs: IN-TF_TAVI_01
Record Dates: First submitted 2020-12-17; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Heart Valve Diseases; Complication,Postoperative
Keywords: length of stay in hospital; transfemoral transaortic valve implantation
MeSH Terms: conditions — Heart Valve Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- analgosedation group: analgosedation concept
- historical group: standard historical concept

SUMMARY:
Transcatheter aortic valve implantation (TAVI) in high-risk patients with severe aortic valve stenosis has developed itself until today as an established minimally invasive alternative procedure worldwide, with a focus on the transfemoral access (TF-TAVI). Meanwhile a number of studies have shown that analgosedation for patients undergoing TF-TAVI is a safe and feasible alternative to general anaesthesia (1). The median length of stay in hospital in Europe is currently 8 days independent to the anesthesia management (2). In the University Hospital Schleswig-Holstein, Campus Kiel, a new TF-TAVI fast-track-concept has been implemented in June 2018. The main intraprocedural aspects of the concept are the preprocedural fluid optimization using transthoracic echocardiography, the idea to decrease or omit the central venous line and the urinary catheter, if reasonable, and finally the individualized low-dose, bolus-based AS.

DETAILED DESCRIPTION:
The investigators are going to monitor 200 patients in 2019 treated with the newly established fast-track concept. During the premedication visit, the investigators informed the patients that the intention is to perform the TF-TAVI, if acceptable, solely in local anaesthesia, in order to minimize potentially adverse pharmacological central effects by analgosedation. After insertion of two peripheral venous lines and an arterial line, monitoring of cerebral oxygenation using near-infrared spectroscopy was established. Transthoracic echocardiography has been performed to evaluate volume status, using the inferior vena cava collapsibility index. Additionally, cardiac output and ejection fraction was calculated.

Based on the data of the investigators and current data from the literature, the investigators assume a postoperative hospital stay of 8 days after TF-TAVI. With a possible reduction of the hospital stay by about 25%, the investigators calculated a case number of 100 patients per group. The study is designed with a control group under standard therapy. Data are recorded and analyzed descriptively. Qualitative comparisons will be made in the discussion of previously published data.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for transfemoral TAVI
* informed written consent

Exclusion Criteria:

* rejection by the patient
* switching to another procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TAVI-patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
length of stay in hospital | through study completion, an average of 1 year
  time in hospital

SECONDARY OUTCOMES:
postoperative complications | through study completion, an average of 1 year
  acute renal failure, pulmonary edema, pneumonia, wound infection
one year mortality | through study completion, an average of 1 year
  survival during one year

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Deutschland (deu), Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renner J, Tesdorpf A, Freitag-Wolf S, Francksen H, Petzina R, Lutter G, Frey N, Frank D. A retrospective study of conscious sedation versus general anaesthesia in patients scheduled for transfemoral aortic valve implantation: A single center experience. Health Sci Rep. 2018 Nov 1;2(1):e95. doi: 10.1002/hsr2.95. eCollection 2019 Jan. PMID 30697594
- [Background] Brecker SJ, Bleiziffer S, Bosmans J, Gerckens U, Tamburino C, Wenaweser P, Linke A; ADVANCE Study Investigators. Impact of Anesthesia Type on Outcomes of Transcatheter Aortic Valve Implantation (from the Multicenter ADVANCE Study). Am J Cardiol. 2016 Apr 15;117(8):1332-8. doi: 10.1016/j.amjcard.2016.01.027. Epub 2016 Jan 28. PMID 26892451